CLINICAL TRIAL: NCT01253213
Title: Exploratory Clinical Trial Using BR55 Targeted Ultrasound Contrast Agent in the Detection of Prostate Cancer by Molecular Imaging of VEGFR2
Brief Title: BR55 in Prostate Cancer: an Exploratory Clinical Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Collaborators: Bracco Imaging S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR55-101
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Ultrasound molecular imaging; Contrast agent; BR55; VEGFR2
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BR55 (Experimental)
  Interventions: Drug: BR55

INTERVENTIONS:
Drug: BR55 — One to two bolus (2nd bolus optional) of BR55 per patient

SUMMARY:
The purpose of this study is to determine whether BR55 is able to identify areas of VEGFR2 expression in human prostate by ultrasound molecular imaging.

This will be compared with histopathology analysis (location based on expression of VEGFR2 in tissue specimens determined by immuno-histochemistry, IHC).

ELIGIBILITY:
Inclusion Criteria:

* Male patient, age ≥ 40 years old
* Has a histology proven focal prostate cancer lesion
* The patient is already scheduled for prostatectomy not earlier than 3 days and at the latest 15 days after BR55 administration
* Provides written Informed Consent and is willing to comply with protocol requirement

Exclusion Criteria:

* Has a body weight greater than 95 kg (this weight limitation is required in order to maintain the active component of the drug under 100μg) according to the indication of the EMEA guideline M3 for this type of study
* Has documented acute prostatitis or urinary tract infections
* Is known to suffer from stable angina pectoris and/or proven coronary disease, or to have symptoms suspicious of coronary disease
* With history of any clinically unstable cardiac condition including class III/IV cardiac failure or right-to-left shunts
* Has had severe cardiac rhythm disorders within the last 7 days
* Has severe pulmonary hypertension (pulmonary artery pressure >90 mmHg) or uncontrolled systemic hypertension or respiratory distress syndrome
* Has received a prostate biopsy procedure within 30 days before admission into this study
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study.
* Is determined by the Investigator that the patient is clinically unsuitable for the study.
* Is incapable of understanding the language in which the information for the patient is given
* Participation in a concurrent clinical trial or in another trial with an investigational compound within the past 30 days;

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
BR55 sensitivity assessment | Day 1
  Assess the ability of BR55 to identify area(s) of VEGFR2 expression in human prostate by ultrasound molecular imaging on the basis of a visual score in comparison with histopathology analysis (location based on expression of VEGFR2 in tissue specimens determined by immuno-histochemistry, IHC).

SECONDARY OUTCOMES:
BR55 specificity assessment | Day 1
  Evaluate the specificity of BR55 targeting for prostate cancer relative to normal prostate gland on the basis of a visual score in comparison with routine histopathology analysis and IHC assessment of VEGFR2 expression in tissue specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Hessel Wijkstra, Dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- AMC University Amsterdam, Amsterdam, Netherlands